CLINICAL TRIAL: NCT03836664
Title: A Randomized, Double-Blinded, Placebo-Controlled, Cross Over Study Evaluating the Efficacy and Safety of Timolol Ophthalmic Solution as an Acute Treatment of Migraine
Brief Title: A Randomized Study Evaluating the Efficacy and Safety of Timolol Ophthalmic Solution as an Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00140465
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Migraine
Keywords: Headache; Acute migraine headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Timolol (Experimental): Participants will be given 0.5% timolol ophthalmic solution to use after migraine onset. Participants will put 2 drops of solution in each eye after migraine and then again 2 hours later.
  Interventions: Drug: Timolol
- Group 2: Placebo (Placebo Comparator): Participants will be given matching placebo (0.9% normal saline solution) to use after migraine onset. Participants will put 2 drops of solution in each eye after migraine and then again 2 hours later.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Timolol — Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
  Other Names: 0.5% timolol ophthalmic solution; beta blocker eye drops
  Arms: Group 1: Timolol
Drug: Placebo — Placebo is normal saline solution that will be supplied in container matched to Timolol container.
  Other Names: inactive drug
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy (headache freedom at 2 hours) of Timolol 0.5% ophthalmic solution compared to placebo in acute treatment of migraine headache. And to assess the safety and tolerability of Timolol 0.5% ophthalmic solution in treatment of acute migraine headache.

DETAILED DESCRIPTION:
Oral beta-blockers are a class of medications frequently used to control blood pressure, angina, and heart irregularities. Certain oral beta-blockers such as propranolol and timolol are used on a daily basis to prevent migraines. However, propranolol and timolol tablets have not been shown to be effective as an acute treatment to stop attacks of migraine because of their longer onset of action. We propose that, since beta-blocker eye drops, unlike tablets are quickly absorbed through the covering of the eye and lining of the nose and can be detected in the bloodstream within minutes, can be beneficial and efficacious in the treatment of headache abortion.

Timolol is a non-selective beta-adrenoreceptor antagonist. Oral timolol (20-30 mg daily) has been studied in 3 randomized controlled trials and have been found to reduce headache frequency by more than 50% when compared to placebo. It has been approved by FDA for prophylactic use in migraine patients and had level A evidence to support this indication. The prophylactic benefit of beta-blockers in migraine treatment is not completely understood. It may be related to the effect of beta-blockers on central autonomic vascular tone center, which in turn modulate the cerebrovascular reactivity to sensory stimulation.Propranolol, a beta-adrenergic blocker modulates serotonergic transmission, regulates peri aqueductal pathway activation and prevents central sensitization, normalizes neuronal excitability in the CNS, and blocks cortical spreading depression (CSD). Topical ocular beta blockers have been reported to be successful in retinal arteriolar spasm, retinal migraines causing visual field defects, migraines causing oculomotor nerve palsy, and as abortive agents in migraine patients. Topical timolol maleate solution 0.5% reaches a concentration of 0.5 ng/ml in the plasma within 4 hours of first dose after being used twice daily for 7 days.

Topical beta-blockers so far have been noted to be effective for acute migraine episodes only in case reports. We believe that this pilot study, to evaluate the efficacy and safety of a timolol eye drop for acute treatment of migraine headaches, will open doors for future trials and larger studies. If successful, this will be able establish the use of beta-blocker eye drops which is a simple, painless and low cost acute treatment of migraine.

The aim of this study is to determine the efficacy of timolol eye drops for the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine, with or without aura, according to ICHD-2 criteria (Appendix A) for at least 1 year prior to screening; experience an average of 1 to 8 migraines per month.
* Females must be practicing an effective method of birth control before entry and throughout the study, or be surgically sterile, or be postmenopausal
* Females of child-bearing potential must have a negative urine pregnancy test
* Subjects should be able to demonstrate the ability to properly administer study medication
* Subjects should be able and willing to read and comprehend written instructions and complete the diary information required by the protocol
* Subjects must be capable, in the opinion of the Investigator, of providing informed consent or assent to participate in the study
* Subjects (and their legally acceptable representatives, if applicable) must provide an informed consent indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Inability to distinguish other headaches from migraine
* Experiences headache of any kind at a frequency greater than or equal to 15 days per month
* Current use of medication for migraine prophylaxis that has not been stable (no dose adjustment) for 30 days prior to screening
* Chronic opioid therapy for headaches (> 3 consecutive days in the 30 days prior to screening)
* Hemiplegic migraine
* History, symptoms or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes
* History of glaucoma and/or current treatment with prescription eye drops
* History of naso-lacrimal duct ("tear duct problem" to patients) obstruction or surgery for such
* Active treatment by ophthalmologist or optometrist for any severe ophthalmic disease or problem
* Any physical problems or co-ordination difficulty or eye avoidance sensitivity ("squeezer") that would preclude proper installation of eye drops in either or both eyes
* History of uncontrolled asthma, COPD, or reversible airway disease which in the opinion of the investigator would be worsened by the use of beta blockers
* History of clinically symptomatic bradycardia, congestive heart failure, or hypotension
* Uncontrolled Diabetes Mellitus
* Uncontrolled Hyperthyroidism
* History (within 2 years) of drug or alcohol abuse
* Systemic disease, which in the opinion of the Investigator, would contraindicate participation
* History of a neurological or psychiatric condition, which in the opinion of the Investigator would contraindicate participation
* History of hypersensitivity or intolerance to beta-blockers eye drops
* Pregnant or lactating women
* Have taken any investigational medication within 12 weeks before randomization, or are scheduled to receive an investigational drug
* Subjects, who in opinion of the Investigator, should not be enrolled in the study because of the precautions, warnings or contra-indications sections of the timolol Package Insert

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dipika Aggarwal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 participants in the age group of 18-65 years were recruited from the general neurology clinics at the University of Kansas Medical Center. One participant did not meet inclusion criteria and was excluded from the study. Finally 25 participants were enrolled. Recruitment period ended from 4/21/17 to 2/23/18.
Pre-assignment Details: Out of the 26 recruited participants, upon screening one participant no more met inclusion criteria due to worsening of his clinical condition. He had an increase in his migraine frequency and therefore, did not meet the inclusion criteria of 1-8 migraine episodes per month. He was considered to be a screen fail and was not enrolled in the study.
Groups:
- Timolol Intervention (2hours), no Washout, Placebo (2 Hours): Participants were randomized to either Timolol/placebo group or placebo/Timolol group.
  Migraine 1: Participants were given 0.5% timolol ophthalmic solution to use after migraine onset. They will put 2 drops of the solution in each eye after migraine onset and again 2 hours later if needed or headache persists.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser
  There was no washout period.
  Migraine 2: Participants were given matching placebo (0.9% normal saline solution) to use after migraine onset. They put 2 drops of solution in each eye after migraine onset and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
- Placebo (2 Hours), no Washout, Timolol (2 Hours): Participants were randomized to either Timolol/placebo group or placebo/Timolol group.
  Migraine 1: Participants were given placebo (0.9% normal saline solution) to use after migraine onset. They put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
  There was no washout period.
  Migraine 2: Participants were given 0.5% timolol ophthalmic solution to use after migraine onset. They put 2 drops of solution in each eye after migraine onset and then again 2 hours later if needed or if headache persisted.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
Period: Overall Study
Arm/Group | Timolol Intervention (2hours), no Washout, Placebo (2 Hours) | Placebo (2 Hours), no Washout, Timolol (2 Hours)
Started | 14 | 11
Completed | 11 | 8
Not Completed | 3 | 3
Not completed — Didn't complete forms and lost drug | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Timolol Intervention (2 Hours), Followed by Placebo (2 Hours): Participants were randomized to either Timolol/placebo group or placebo/Timolol group.
  Migraine 1: Participants were given 0.5% timolol ophthalmic solution to use after migraine onset. They will put 2 drops of the solution in each eye after migraine onset and again 2 hours later if needed or headache persists.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser
  There was no washout period.
  Migraine 2: Participants were given matching placebo (0.9% normal saline solution) to use after migraine onset. They put 2 drops of solution in each eye after migraine onset and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
- Placebo (2 Hours), Followed by Timolol Intervention (2 Hours): Participants were randomized to either Timolol/placebo group or placebo/Timolol group.
  Migraine 1: Participants were given matching placebo (0.9% normal saline solution) to use after migraine onset. They put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
  There was no washout period.
  Migraine 2: Participants were given 0.5% timolol ophthalmic solution to use after migraine onset. They put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
- Total: Total of all reporting groups
Arm/Group | Timolol Intervention (2 Hours), Followed by Placebo (2 Hours) | Placebo (2 Hours), Followed by Timolol Intervention (2 Hours) | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Headache Severity
Description: Measure of the change in severity using visual analogue pain scale ranging from 0-10 with zero being no pain and ten being worst pain. Scale will be completed after each migraine episode over course of participation in study, up to 8 weeks.
Time Frame: Headache/ pain severity at onset and at 120 minutes post intervention use
Population: All participants
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- All Participants Post Timolol: Participants given 0.5% timolol ophthalmic solution to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
- All Participants Post Placebo: Participants given matching placebo (0.9% normal saline solution) to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
Arm/Group | All Participants Post Timolol | All Participants Post Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 2.00 [1.04 to 2.96] | 2.00 [0.72 to 3.07]

2. Secondary Outcome: Adverse Reaction From Using Timolol Eye Drops
Description: Measured by number of adverse events experienced by the participants from the intervention. Each adverse event was counted as one.
Time Frame: 8 weeks
Population: total number of adverse events in each group
Measure: Number; unit: events
Groups:
- Total Number of Adverse Events Post Timolol Intervention: Participants given 0.5% timolol ophthalmic solution to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
- Total Number of Adverse Events Post Placebo: Participants given matching placebo (0.9% normal saline solution) to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
Arm/Group | Total Number of Adverse Events Post Timolol Intervention | Total Number of Adverse Events Post Placebo
Number analyzed (Participants) | 19 | 19
events | 2 | 3

3. Secondary Outcome: Number of Participants Satisfied With Intervention
Description: Measured by patient-reported satisfaction questionnaire. Satisfaction level was looked at as "satisfactory and very satisfactory" compared to "neutral and unsatisfied".
Time Frame: 8 weeks
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants Satisfied Post Timolol Intervention: Participants given 0.5% timolol ophthalmic solution to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
- Number of Participants Satisfied Post Placebo: Participants given matching placebo (0.9% normal saline solution) to use after migraine onset. Participants put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or if headache persisted.
  Placebo: Placebo is normal saline solution supplied in container matched to Timolol container.
Arm/Group | Number of Participants Satisfied Post Timolol Intervention | Number of Participants Satisfied Post Placebo
Number analyzed (Participants) | 19 | 19
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected within 1 day of drug administration. All participants were advised to report any adverse event within 24 hours.
Description: Participants were advised to call with minor side effects/ adverse events within 24 hours, and go to nearest ER in case of any serious adverse event.
Groups:
- All Participants Post Timolol: Participants will be given 0.5% timolol ophthalmic solution to use after migraine onset. Participants will put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or headache persists.
  Timolol: Timolol is a clear solution supplied in a plastic ophthalmic dispenser.
- All Participants Post Placebo: Participants will be given matching placebo (0.9% normal saline solution) to use after migraine onset. Participants will put 2 drops of solution in each eye after migraine and then again 2 hours later if needed or headache persists.
  Placebo: Placebo is normal saline solution that will be supplied in container matched to Timolol container.
Arm/Group | All Participants Post Timolol | All Participants Post Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Post Timolol (N=19) | All Participants Post Placebo (N=19)
Eyes burning/ stinging (Eye disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Participant compliance was also found to be a big limitation with 6 participants considered as study drop outs since they did not return study drug/ forms even after repeated attempts to contact them. This led to loss of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03836664/Prot_SAP_000.pdf